CLINICAL TRIAL: NCT01898637
Title: A Simple Clinical Tool to Help Diagnose Pulmonary Embolism: Phase 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Scott Keller, PI, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-009527
Record Dates: First submitted 2013-06-28; First posted 2013-07-12 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; pulse oximetry; change in oxygen saturation; hypoxemia; emergency department; deep inspiration; vital capacity; clinical diagnosis
MeSH Terms: conditions — Pulmonary Embolism; Hypoxia; Emergencies

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proven pulmonary embolism. (Active Comparator): Augmented pulse oximetry using incentive spirometer. Emergency Department patients with pulmonary embolism.
  Interventions: Other: Augmented pulse oximetry using incentive spirometer.; Device: Incentive spirometer.
- Control patients (Other): Augmented pulse oximetry using incentive spirometer. Emergency Department patients who do not have pulmonary embolism.
  Interventions: Other: Augmented pulse oximetry using incentive spirometer.; Device: Incentive spirometer.

INTERVENTIONS:
Other: Augmented pulse oximetry using incentive spirometer. — Augmented pulse oximetry using incentive spirometer.
Device: Incentive spirometer. — The incentive spirometer is a simple passive device that measures the amount of air a person can inhale.
  Other Names: AirLife Volumetric Incentive Spirometer.

SUMMARY:
The goal of this project is to determine if the change in oxygen saturation during deep inspiration ("augmented pulse oximetry") can be used as a method to rule out pulmonary embolism (PE). The investigators propose to evaluate a simple, non-invasive clinical tool to help rule out PE. The investigators plan to measure the oxygen saturation of 40 consecutive patients with newly-diagnosed PE (within 60 minutes of diagnosis) and 80 matched controls who do not have a PE. Trained, blinded Respiratory Therapists or Study Coordinators will record each patient's oxygen saturation before, during, and after a 2-minute period of deep inspirations (vital capacity [the maximal amount of air that can be inhaled, measured in milliliters]) using an incentive spirometer. The investigators' central hypothesis is that persons with a PE will not respond to augmented pulse oximetry and will not significantly improve or normalize their oxygen saturation.

DETAILED DESCRIPTION:
Patients will be identified and enrolled by the Mayo Clinic St. Marys Emergency Department staff as they are undergoing medical care in the Emergency Department.

The investigators will calculate the difference in oxygen saturation pre- and post-deep inspiration (ΔSpO2 at 1 minute, 2 minutes and 4 minutes), and then correlate these values with the CT result.

In cases of PE, The investigators expect the SpO2 to remain unchanged, or to change less than 3-5%. The investigators expect alternate hypoxemic conditions to have a significantly greater increase in SpO2.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater.
* Agrees and able to participate in the study.
* Room air SpO2 (oxygen saturation) less than 92% and newly-diagnosed PE (or controls with no PE) based on CT angiogram result.

Exclusion Criteria:

* Clinical concern for instability.
* Systolic blood pressure less than 100 mm Hg.
* Heart rate ≥140 beats per minute.
* Oxygen saturation less than 85% with more than 4 L supplemental oxygen.
* Unable to participate/comply with instructions for using the incentive spirometer.
* Patients from the Federal Medical Center in Rochester, Minnesota.
* Patients who do not speak English (due to the need for expediency).

Patients will be under the care of the Emergency Department team who have the skills and resources to monitor and treat patients if they were to become unstable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-06; Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Change in oxygen saturation using augmented pulse oximetry for patients with and without pulmonary embolism. | Oxygen saturation (SpO2) will be recorded prior to using the spirometer, at 1 minute (during use of the spirometer), at 2 minutes (at the end of using the spirometer), and at 4 minutes.
  Trained, blinded Respiratory Therapists or Study Coordinators will record each patient's oxygen saturation before, during, and after a 2-minute period of deep inspirations (vital capacity) using an incentive spirometer. The investigators will calculate the difference in oxygen saturation pre- and post-deep inspiration (ΔSpO2 at 1 minute, 2 minutes and 4 minutes), and then correlate these values with the CT result.

SECONDARY OUTCOMES:
Vital capacity (the maximal amount of air that can be inhaled, measured in milliliters) during augmented pulse oximetry. | The single maximum value obtained prior to using the spirometer, at 1 minute (during use of the spirometer), at 2 minutes (at the end of using the spirometer), and at 4 minutes.
  The single maximum value obtained before, during, or after use of the incentive spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: A. S. Keller, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials